CLINICAL TRIAL: NCT01518855
Title: Clinical Effect and Cost Effectiveness of Ca Antagonist in Combination With AII Receptor Antagonist in Patient With Essential Hypertension (PMS Study)
Brief Title: Controlled Release Nifedipine and Valsartan Combination Therapy in Patients With Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Medical Development Japan, Bayer Yakuhin Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11518
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nifedipine; Amlodipine; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Adalat CR 20-40mg od + Diovan 40-80mg od
  Interventions: Drug: Nifedipine (Adalat, BAYA1040); Drug: Diovan
- Arm 2 (Active Comparator): Norvasc 2.5-5mg od + Diovan 40-80mg od
  Interventions: Drug: Amlodipine (Norvasc); Drug: Diovan

INTERVENTIONS:
Drug: Nifedipine (Adalat, BAYA1040)
  Arms: Arm 1
Drug: Amlodipine (Norvasc)
  Arms: Arm 2
Drug: Diovan

SUMMARY:
The primary objective of this study is to investigate incremental cost effectiveness of Nifedipine CR and Amlodipine in combination therapy with Valsartan for the treatment of essential hypertensive patients.

To investigate incremental cost effectiveness, primary variables are mean treatment cost and achievement rate to target blood pressure level at the end of double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

Untreated patients or patients with previous treatment by antihypertensive agents whose blood pressure at sitting position at the time of the entry (Visit 1) is:

* SBP>/=160mmHg or DBP>/=100mmHg for untreated patients (SBP Systolic blood pressure, DBP Diastolic blood pressure)
* SBP>/=150mmHg or DBP>/=95mmHg for patients with previous treatment by antihypertensive agents

Exclusion Criteria:

* Patients whose blood pressure on either day of Visit 1 or 2 is: SBP > 200mmHg or DBP > 120mmHg.
* Patients with secondary hypertension or hypertensive emergency such as malignant hypertension.
* Patients with a history of cardiovascular or cerebrovascular ischemic event (stroke, transient ischemic attack, myocardial infarction or unstable angina) within six months prior to the study.
* Patients with a history of intracranial or subarachnoid hemorrhage within six months prior to the study.
* Patients with uncontrolled diabetes (HbA1c >/=8%)
* Patients with bradycardia or tachycardia (<50 bpm, >/=100 bpm), arrhythmia such as atrioventricular block (second and third degree), sinoatrial block or atrial fibrillation.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2004-03; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Mean treatment cost* for 16-week of double-blind treatment period | 16 weeks
  * Including treatment cost for the drug related AEs. The sponsor will calculate the cost based on the tariff of health insurance scores.
Proportion of participants** achieving target blood pressure at the end of double-blind treatment period | at week 16
  **For subjects aged under 60 years: SBP<130mmHg and DBP<85mmHg, for subjects aged 60 years or over: SBP<140mmHg and DBP<90mmHg (SBP Systolic blood pressure, DBP Diastolic blood pressure)

SECONDARY OUTCOMES:
Treatment cost per subject to achieve the target blood pressure (Total costs for the double-blind treatment period / Number of patients who achieve the target blood pressure at the end of double-blind treatment period) | 16 weeks
The change in blood pressure (SBP and DBP) from the baseline (end of pretreatment period) . | baseline to week 16
Proportion of participants for each age group to target blood pressure level | at week 16
Incidence of treatment-emergent drug-related adverse events | 16 weeks
Safety variables will be summarized using descriptive statistics based on adverse events collections | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Japan (4):
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Setagaya-ku, Tokyo
  - Shinjuku-ku, Tokyo